CLINICAL TRIAL: NCT05535075
Title: Impact of Model-informed Precision Dosing of Vancomycin in Adults: a Randomized, Clinical Trial
Brief Title: Model-informed Precision Dosing of Vancomycin in Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC-10433; 2021-003670-31 (EudraCT Number)
Record Dates: First submitted 2022-05-13; First posted 2022-09-10 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Vancomycin
Keywords: vancomycin; model-informed precision dosing; dose calculator; non-critically ill adults
MeSH Terms: interventions — Vancomycin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and legal representatives are blinded for the allocation to the intervention or standard-of-care arm until the end of study. The statistician is kept blinded until after data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Vancomycin treatment (Active Comparator): Vancomycin standard-of-care dosing and therapeutic drug monitoring (TDM), according to institutional guidelines during 20 day study period
  Interventions: Drug: Vancomycin
- Vancomycin model-informed precision dosing (Experimental): Area Under the Concentration-time curve ((AUC)/Minimal Inhibitory Concentration (MIC)-based model-informed precision dosing of vancomycin using a dosing calculator during 20 day study period
  Interventions: Device: Vancomycin model-informed precision dosing; Drug: Vancomycin

INTERVENTIONS:
Device: Vancomycin model-informed precision dosing — A dosing calculator is used for a posteriori calculation of vancomycin dose using a target AUC/MIC between 400-600 mg*h/L
  Other Names: Dosing calculator
  Arms: Vancomycin model-informed precision dosing
Drug: Vancomycin — Vancomycin treatment
  Other Names: Vancomycin treatment

SUMMARY:
The overall objective of this project is to investigate the utility of model-informed precision dosing (MIPD) of vancomycin in non-critically ill adults. This evaluation includes a comparison with the more standard approach on clinical and patient-oriented measures.

DETAILED DESCRIPTION:
Vancomycin is an antibiotic with a narrow therapeutic-toxic margin. This means that the minimum and maximum target blood target levels differ little from each other. Too low concentrations will reduce the effect of the antibiotic; higher concentrations may result in serious side effects, including renal toxicity. Vancomycin dosing tailored to the individual patient is challenging.

Currently, the vancomycin dose is adjusted based on a measured vancomycin blood concentration (if too high or too low). Despite this measurement, quickly achieving target concentrations remains a major challenge.

This multicenter, individual randomized study investigates the added value of a user-friendly computer program for calculating the vancomycin dose in non-critically ill adults, compared to the current standard-of-care. Specifically, the investigators will study whether the use of this computer program leads to a shorter time to reach target concentrations, a reduction in the number and severity of side effects on the kidney and a reduction in patient burden.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* admitted to a participating ward unit
* a suspected or confirmed Gram positive infection
* planned to start of started on intravenous continuous infusion vancomycin treatment
* participant or legal representative signed the informed consent form
* not previously enrolled in this trial

Exclusion Criteria:

* serum creatinine level at inclusion is above 2.5 mg/dL
* undergoing extracorporeal treatment at inclusion (e.g. extracorporeal membrane oxygenation, dialysis, body cooling)
* patient death is deemed imminent and inevitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reaching target 24h AUC/MIC | 48 to 72 hours after start vancomycin treatment
  Therapeutic AUC/MIC target range is 400-600

SECONDARY OUTCOMES:
Proportion of patients with (worsening) acute kidney injury (AKI) during vancomycin treatment | From start date of vancomycin treatment until stop date vancomycin treatment or study day 20, whichever comes first
  AKI categories are defined according to the Kidney Disease Improving Global Outcomes (KDIGO) criteria from stage 1 to 3 (worst)
Proportion of patients reaching target 24h AUC/MIC | 72 to 96 hours after start vancomycin treatment
  Therapeutic AUC/MIC target range is 400-600
Proportion of time within therapeutic target | From start date of vancomycin treatment until stop date vancomycin treatment or study day 20, whichever comes first
  Therapeutic AUC/MIC target range is 400-600

OTHER OUTCOMES:
Number of (additional) blood samples to first target attainment during vancomycin treatment | From start date of vancomycin treatment until date of first vancomycin target attainment or study day 20, whichever comes first
  An additional blood sample is defined as a sample for vancomycin TDM taken at another timepoint of routine biochemical monitoring samples.
Cumulative number of (additional) blood samples | From start date of vancomycin treatment until stop date vancomycin treatment or study day 20, whichever comes first
  An additional blood sample is defined as a sample for vancomycin TDM taken at another timepoint of routine biochemical monitoring samples.
Number of dose adjustments to first target attainment | From start date of vancomycin treatment until date of first vancomycin target attainment or study day 20, whichever comes first
  Target in Model-Informed Precision Dosing arm: 24h AUC/MIC : 400-600; in comparator arm: target concentration range according to institutional guidelines
Cumulative vancomycin dose | From start date of vancomycin treatment until stop date vancomycin treatment or study day 20, whichever comes first
  Total cumulative exposure (AUC) during treatment
Cumulative vancomycin AUC | From start date of vancomycin treatment until stop date vancomycin treatment or study day 20, whichever comes first
  Total exposure (AUC) during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Pieter De Cock, Prof, Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - General Hospital Sint-Jan Brugge, Bruges
  - Ghent University Hospital, Ghent